CLINICAL TRIAL: NCT07245004
Title: The Effect of Cryotherapy on Postoperative Pain for Pulpotomy in Permanent Mature Carious Posterior Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Effect of Cryotherapy on Postoperative Pain for Pulpotomy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sirawut Hiran-us (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Sponsor-Investigator, Sirawut Hiran-us, Associate Professor, Chulalongkorn University
Organization: Chulalongkorn University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBC 32/2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pulpitis - Irreversible
Keywords: Pulpotomy; Cryotherapy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Addition of Cryotherapy on pulpotomy (Experimental): After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the refrigerator set to 2.5°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion: 5 ml in each of 4 syringes, administered every 1.25 minutes per syringe.
  Interventions: Other: Cryotherapy
- Rountine pulpotomy (No Intervention): After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the room temperature 25°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion.

INTERVENTIONS:
Other: Cryotherapy — After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the refrigerator set to 2.5°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion: 5 ml in each of 4 syringes, administered every 1.25 minutes per syringe.
  Arms: Addition of Cryotherapy on pulpotomy

SUMMARY:
The goal of this clinical trial is to investigate the effect of cryotherapy on post-operative pain for pulpotomny in permanent mature carious posterior teeth with symptomatic irreversible pulpitis. The main question is: Do cryotherapy reduce post-operative pain and improve QoL in interested samples?

[primary hypothesis or outcome measure 1] Post-operative pain by Numerical rating scale scores.

[primary hypothesis or outcome measure 2] QoL of patients by OHIP-14

If there is a comparison group: Researchers will compare pulpotomy incorperated with cryotherapy and without.

Participants will scoring VAS scores and OHIP-14 before and after treatment at designated time points.

DETAILED DESCRIPTION:
Materials and methods Study design and setting This study is a prospective, single-center, double-blinded, parallel-group, randomized controlled trial conducted at the Dental Department, Yala Hospital. All clinical procedures are performed by a single trained operator.

Study participants Inclusion Criteria

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent posterior teeth diagnose with symptomatic irreversible pulpitis. Diagnoses are confirmed using Electric Pulp Test(EPT) and cold test. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013).
* Posterior teeth with moderate or severe pain according to the Numerical rating scale (NRS):no pain(0), mild pain, non-disruptive to routine activity (1-3), moderate pain, interferes with daily life but no need analgesic intake (4-6) and severe pain, interferes with daily life and need analgesic intake (7-10).
* Teeth that response negatively to percussion and palpation tests.
* Teeth without periapical pathosis.
* Teeth are restorable with direct composite restoration. Exclusion Criteria
* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Patients who had taken analgesics or anti-inflammatory drugs within the previous 24 hours.
* Patients taking opioids.
* Known allergies to non-steroidal anti-inflammatory drugs (NSAIDs).
* Pregnant or lactating patients.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening.
* Bleed cannot be stopped within 8 minutes after full pulpotomy26,27 Treatment procedure A comprehensive medical and dental history is taken before treatment. Preoperative data, including age, sex, tooth number, and pain intensity are recorded in a predesigned patient's chart. The severity of pain is measured using VAS 0-10. The treatment, the study design, alternative treatment modalities, potential benefits, risks, and follow-up protocol are explained to the qualifying patients and informed consent is obtained from the voluntary patients who are willing to participate in the study.

Sample size calculation The sample size calculation was based on a study by Kubra G. and Koray Y. 202539 using a G*Power v.3.1 (Heinrich Heine, Dusseldorf University, Dusseldorf Germany) with a 95% power, a 5% α error, and an effect size of 0.75. The minimum sample size was calculated to be 78. Considering patients lost to follow-up, a total of 82 teeth from different patients are included in this study.

Randomization and masking Block randomization with variable 4 block sizes is used to generate a sequence of random numbers for allocating the patients equally into two study groups. Each random blocks are sealed in an opaque envelope which is opened at the beginning of the clinical trial by dental assistant who the one only know the intervention and prepare the intervention for operator. New block will be open after all the patients in the previous block was completed and repeat until the end of the clinical trials to ensure the equality of group distribution: The VTP with and without cryotherapy intervention groups.

Intervention

All the treatment is carried out by a single operator under magnification(3x loupes) and illumination. All the patients received a topical anesthesia before local anesthesia. An inferior alveolar nerve block (1.8 ml 2% Lidocaine with epinephrine 1:100,000) + buccal infiltration (1.7 ml 4% Articaine with epinephrine 1:100,000) for mandibular teeth, buccal infiltration (1.8 ml 2% Lidocaine with epinephrine 1:100,000) for maxillary teeth. The anesthesia is confirmed by negative response to EPT. The pulpotomy procedure is performed under rubber dam isolation in a single visit. If the patient experienced pain during the procedure, an additional anesthesia is used to achieve profound pulpal anesthesia by intraligament injection with 0.3 ml 2% Lidocaine with epinephrine 1:100,000. The operating field is disinfected with iodine and alcohol. A high-speed diamond airotor operates under air water coolant to outline the cavity. Low speed round steel bur and a spoon excavator are used to remove the soft carious dentine using nonselective caries removal from the periphery towards the centre of the carious lesion. The deepest layer of carious dentine is thereafter disinfected with 2 ml of 2.5% NaOCl prior to pulpal exposure. The new high-speed sterile diamond airotor is used to completely remove the coronal pulp tissue. Then rinse with of 2.5% NaOCl solution up to 8 minutes to arrest the bleeding. The time to achieve hemostasis is recorded in minutes and seconds. The diagnosis of vital inflamed pulp is confirmed by the presence of bleeding in the pulp chamber. The dental assistant will bring an insulated syringe containing different intervention as follow:

Group I (Cryotherapy): After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the refrigerator set to 2.5°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion: 5 ml in each of 4 syringes, administered every 1.25 minutes per syringe.

Group II (Control): After hemostasis is achieved, the pulpotomy area is irrigated for 5 minutes with normal saline solution, which is kept in the room temperature 25°C (measuring with thermometer and record) by using a disposable insulated 5 ml syringe and 21-gauge needle is placed 1-2 mm above the root canal orifices and is constantly moved in a circular motion.

In both study groups, 2 mm calcium silicate cement putty type (TFRRM) is placed as a capping agent over the residual pulp. The tooth is restored with Resin Modified Glass Ionomer Cement (RMGIC) base (Vitrebond, 3M) and composite restoration (Z350XT, 3M) and polishing in the same visit.

The full pulpotomy cases where bleeding from residual pulp cannot be arrested within 8 minutes, are excluded from the study, and pulpectomy are performed. Immediate post-operative periapical radiograph is taken.

Post-operative evaluation The patient's postoperative pain score and frequency of analgesic intake are recorded by calling and asking for information during at 6, 24, 48, and 72 hours. Ibuprofen 400 mg 10 tablets and Paracetamol 500 mg 10 tablets will be prescribed for every patient in advance.

If patients have a complaint of pain, they can have 1 tablet of ibuprofen 400 mg, with a note down the number and time of intake. If the patient can't tolerate the pain after taken 1 tablet of ibuprofen for 60 minutes, there can have another 1 tablet of paracetamol, with a note down the number and time of intake. Patients are also informed to return to the clinician in case of persistent severe pain in the post-intervention period, even after taking prescribed medication.

Patient will be asked to complete the OHIP-14 survey before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent posterior teeth diagnose with symptomatic irreversible pulpitis. Diagnoses are confirmed using Electric Pulp Test(EPT) and cold test. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013).
* Posterior teeth with moderate or severe pain according to the Visual Analog Scale(VAS):no pain(0), mild pain, non-disruptive to routine activity (1-3), moderate pain, interferes with daily life but no need analgesic intake (4-6) and severe pain, interferes with daily life and need analgesic intake (7-10).
* Teeth that response negatively to percussion and palpation tests.
* Teeth without periapical pathosis.
* Teeth are restorable with direct composite restoration.

Exclusion Criteria:

* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Patients who had taken analgesics or anti-inflammatory drugs within the previous 24 hours.
* Patients taking opioids.
* Known allergies to non-steroidal anti-inflammatory drugs (NSAIDs).
* Pregnant or lactating patients.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening.
* Bleed cannot be stopped within 8 minutes after full pulpotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score | 6, 24, 48, 72, 96, 120, 148, 172, 196 hours after treatment
  Pain was recorded using a numerical rating scale (NRS) which minimum is 0 and maximum is 10. Higher scores indicate worse pain, while lower scores indicate better outcomes.

SECONDARY OUTCOMES:
Patient quality of life | Before treatment and at 7 days after treatment
  Assessment of quality of life of patient before and after treatment using OHIP-14 questionaire.
  The minimum score is 14 maximum is 70. Higher score mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sirawut Hiran-us, DDS, MSc, High Grad Dip, FRCDS, Study Director — Faculty of Dentistry, Chulalongkorn University; Sawat Pojlerdarun, DDS, Higher Grad Dip, FRCDS, Principal Investigator — Dental Department, Yala Hospital
Locations (1):
- Yala Hospital, Yala, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gurler K, Yilmaz K. The Effect of Novel Cryotherapy Technique on Postoperative Pain for Pulpotomy in Permanent Molars with Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial. J Endod. 2025 May;51(5):547-553. doi: 10.1016/j.joen.2025.01.020. Epub 2025 Feb 3. PMID 39909197